CLINICAL TRIAL: NCT04236830
Title: Effectiveness of Silver Diamine Fluoride/ Potassium Iodide in Indirect Pulp Capping of Young Permanent Molars (a Randomized Controlled Clinical Trial)
Brief Title: Silver Diamine Fluoride/ Potassium Iodide in Indirect Pulp Capping of Young Permanent Molars
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Dental Public Health clinical instructor and study statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDF/potassium iodide
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Tertiary Dentine; Indirect Pulp Capping
Keywords: Silver diamine fluoride/ potassium iodide; glass ionomer cement
MeSH Terms: conditions — Dentin, Secondary | interventions — silver diamine fluoride; Potassium Iodide

STUDY DESIGN:
Intervention Model Description: This is a 3 arm clinical trial. All selected first permanent molars will be randomly equally allocated into three groups according to capping material used.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of examiners is impossible to be done during intervention and follow up due to different natures of the materials. However, participants and outcome assessors could be blinded (double blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silver diamine fluoride/ potassium iodide group (Experimental): Riva Star Silver diamine fluoride 38% and potassium iodide, SDI, Bayswater, Australia
  Interventions: Drug: Silver diamine fluoride/ potassium iodide
- Silver diamine fluoride group (Experimental): Advantage arrest TM, Elevate Oral Care, USA
  Interventions: Drug: Silver diamine fluoride
- Resin modified glass ionomer cement group (Active Comparator): Riva light cure, SDI, Bayswater, Australia
  Interventions: Drug: Resin modified glass ionomer cement

INTERVENTIONS:
Drug: Silver diamine fluoride/ potassium iodide — Thirty six first permanent molars will receive 38% SDF/KI as an indirect pulp capping material.
  Other Names: SDF/KI
  Arms: Silver diamine fluoride/ potassium iodide group
Drug: Silver diamine fluoride — Thirty six first permanent molars will receive 38% SDF as an indirect pulp capping material.
  Other Names: SDF
  Arms: Silver diamine fluoride group
Drug: Resin modified glass ionomer cement — Thirty six first permanent molars will receive RMGIC as an indirect pulp capping material.
  Other Names: RMGIC
  Arms: Resin modified glass ionomer cement group

SUMMARY:
The aim of this study is to evaluate and compare the clinical effectiveness of 38% silver diamine fluoride with and without potassium iodide with that of resin modified glass ionomer cement in indirect pulp capping of young permanent molars.

DETAILED DESCRIPTION:
A sample of children with an age range of 6-9 years, having a first permanent molar erupted with deep occlusal carious lesion, will be selected from the outpatient clinic of Pediatric Dentistry and Public Health Department, Faculty of Dentistry, Alexandria University after securing necessary consents. All selected 108 first permanent molars will be randomly equally allocated into three groups according to capping material used. Group I (n=36) SDF/ KI and Group II (n=36) SDF and Group III (n=36) Glass ionomer cement. Indirect pulp capping treatment procedure will be performed with identical protocols except for the capping material to be used and its application will be according to manufacturer's instructions. Glass ionomer cement will be used as a base and resin-based composite restoration will be used in the three groups.

ELIGIBILITY:
Inclusion Criteria:

For children:

1. Children who are generally healthy.
2. Children having a deep dentin carious lesion in a permanent first molar (upper or lower).
3. Parents signed informed consent.

For first permanent molars:

1. Cavitated class I carious lesions with opaque or discolored enamel exposing the dentin beneath corresponding to ICDAS II score 5 and 6 (visible dentin). (Ekstrand KR, Martignon S, Ricketts D, Qvist V. 2007)
2. Teeth having lesions that are considered active according to ICDAS II activity criteria for primary coronal caries. (Ekstrand KR, Martignon S, Ricketts D, Qvist V. 2007; Dikmen B. 2015)
3. Immature with open apex as revealed by periapical X-ray.

Exclusion Criteria:

For children:

1. Any allergy reported by the parents. (Crystal YO, Marghalani AA, Ureles SD, Wright JT, Sulyanto R, Divaris K, et al. 2017)
2. Children unable to return for recall visits.

For first permanent molars:

1. Any clinical signs of irreversible pulpitis (spontaneous pain, pain on percussion, abscess, sinus.
2. Any radiographic sign of irreversible pulp pathologies or necrosis periapical radiolucency, internal or external root resorption).
3. Teeth with inactive lesions. (Ekstrand KR, Martignon S, Ricketts D, Qvist V. 2007; Dikmen B. 2015)

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 6 months
  Postoperative pain will be assessed by questioning the patient or the guardian whether there is postoperative pain or not, Binary (yes or no). (American Academy of Pediatric Dentistry. 2019)
Postoperative pain | 12 months
  Postoperative pain will be assessed by questioning the patient or the guardian whether there is postoperative pain or not, Binary (yes or no). (American Academy of Pediatric Dentistry. 2019)
Tooth Vitality | 6 months
  Tooth vitality will be assessed by vitality test using thermal stimulation, binary (yes or no). (American Academy of Pediatric Dentistry. 2019)
Tooth Vitality | 12 months
  Tooth vitality will be assessed by vitality test using thermal stimulation, binary (yes or no). (American Academy of Pediatric Dentistry. 2019)
Success of the restoration | 6 months
  Clinical success of the whole restoration will be ranked according to Modified Ryge/USPHS Clinical Criteria (Colour, marginal adaptability, marginal staining, and secondary caries). (Moncada G, Silva F, Angel P, Oliveira Jr O, Fresno MC, Cisternas P, et al. 2014)
Success of the restoration | 12 months
  Clinical success of the whole restoration will be ranked according to Modified Ryge/USPHS Clinical Criteria (Colour, marginal adaptability, marginal staining, and secondary caries). (Moncada G, Silva F, Angel P, Oliveira Jr O, Fresno MC, Cisternas P, et al. 2014)
Radiographic evaluation or root lengthening | 6 months
  Root lengthening will be assessed by measuring the root length in mm from cement-enamel junction on standardized digital radiographs taken by parallel technique (digora software). (Flake NM, Gibbs JL, Khan AA. 2014)
Radiographic evaluation or root lengthening | 12 months
  Root lengthening will be assessed by measuring the root length in mm from cement-enamel junction on standardized digital radiographs taken by parallel technique (digora software). (Flake NM, Gibbs JL, Khan AA. 2014)
Radiographic evaluation of reparative dentin formation | 6 months
  Reparative dentin formation, if present, will be measured in millimetre on standardized digital radiographs taken by parallel technique (digora software). (Menon NP, Varma BR, Janardhanan S, Kumaran P, Xavier AM, 2016)
Radiographic evaluation of reparative dentin formation | 12 months
  Reparative dentin formation, if present, will be measured in millimetre on standardized digital radiographs taken by parallel technique (digora software). (Menon NP, Varma BR, Janardhanan S, Kumaran P, Xavier AM, 2016)
Radiographic evaluation of reparative dentin volume | 12 months
  This was measured using cone beam computed Tomography (CBCT). Reparative dentin radiodensity will be measured in Hounsfield units (HU). (Mathur VP, Dhillon JK, Logani A, Kalra G. 2016)

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Baraka, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Magda El-Tekeya, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Niveen Bakry, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Fontana Margherita, Study Chair — University of Michigan
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Ekstrand KR, Martignon S, Ricketts DJ, Qvist V. Detection and activity assessment of primary coronal caries lesions: a methodologic study. Oper Dent. 2007 May-Jun;32(3):225-35. doi: 10.2341/06-63. PMID 17555173
- [Background] Dikmen B. Icdas II criteria (international caries detection and assessment system). J Istanb Univ Fac Dent. 2015 Oct 21;49(3):63-72. doi: 10.17096/jiufd.38691. eCollection 2015. PMID 28955548
- [Background] Crystal YO, Marghalani AA, Ureles SD, Wright JT, Sulyanto R, Divaris K, Fontana M, Graham L. Use of Silver Diamine Fluoride for Dental Caries Management in Children and Adolescents, Including Those with Special Health Care Needs. Pediatr Dent. 2017 Sep 15;39(5):135-145. PMID 29070149
- [Background] Guideline on Pulp Therapy for Primary and Immature Permanent Teeth. Pediatr Dent. 2016 Oct;38(6):280-288. No abstract available. PMID 27931467
- [Derived] Baraka MMAL, Cevidanes L, Tekeya M, Bakry N, Ruellas A, Botero T, Benavides E, Fontana M. Three-Dimensional Assessment of Radiographic Changes after Indirect Pulp Capping Using Silver Diamine Fluoride with or without Potassium Iodide in Young Permanent Teeth (12-Month RCT). Caries Res. 2023;57(2):177-188. doi: 10.1159/000529893. Epub 2023 Mar 6. PMID 36878216
- [Derived] Baraka M, Tekeya M, Bakry NS, Fontana M. Twelve-month randomized controlled trial of 38% silver diamine fluoride with or without potassium iodide in indirect pulp capping of young permanent molars. J Am Dent Assoc. 2022 Dec;153(12):1121-1133.e1. doi: 10.1016/j.adaj.2022.08.008. Epub 2022 Oct 15. PMID 36253166